CLINICAL TRIAL: NCT03458143
Title: Study of Respiratory Depression During Analgosedation Technique Combining Remifentanyl and Ketamine in TCI for Oocyte Retrieval
Brief Title: Respiratory Depression During an Analgosedation Combining Remifentanil and Ketamine in TCI for Oocyte Retrieval
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Luc Barvais, MD PhD, Erasme University Hospital
Other Study IDs: P2018/016
Record Dates: First submitted 2018-02-14; First posted 2018-03-08 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Oocyte Retrieval; Sedation, Conscious; Ventilatory Depression
Keywords: ketamine; remifentanil
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Ketamine; Conscious Sedation; Remifentanil; Oocyte Retrieval

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma/Serum for Ketamine dosage after the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ketamine 150 ng/ml: The first group will receive the classical premedication with 2 mg of Midazolam. A bolus dose of Ketamine will be given, then to be titrated in TCI mode with a target concentration of 150 ng/ml. Right after, the Remifentanil TCI will be started at a concentration of 1 ng/ml and the procedure can begin.
  Interventions: Drug: Ketamine 150 ng/ml; Drug: Remifentanil; Procedure: Oocyte retrieval
- ketamine 200 ng/ml: The second group will be treated in the exact way as the first, with the exception that the target effect site concentration is aimed at 200 ng/ml.
  Interventions: Drug: Remifentanil; Procedure: Oocyte retrieval; Drug: Ketamine 200 ng/ml

INTERVENTIONS:
Drug: Ketamine 150 ng/ml — conscious sedation in TCI-mode
  Other Names: conscious sedation
  Groups: ketamine 150 ng/ml
Drug: Remifentanil — conscious sedation in TCI-mode
  Other Names: conscious sedation
Procedure: Oocyte retrieval — Oocyte retrieval for In Vitro Fertilization
Drug: Ketamine 200 ng/ml — conscious sedation in TCI-mode
  Other Names: conscious sedation
  Groups: ketamine 200 ng/ml

SUMMARY:
This study evaluates the effect of the addition of ketamine to a conscious sedation protocol including remifentanil during oocyte retrieval. The investigators will have 2 groups with different target effect site concentrations, namely 150 ng/ml and 200 ng/ml.

DETAILED DESCRIPTION:
The actual protocol for conscious sedation during oocyte retrieval in at the Erasmus hospital (Brussels) consists of Remifentanil in TCI-mode, with premedication by Midazolam. However, episodes of bradypnaea with or without desaturation are still common.

The primary objective is to observe if with the addition of ketamine, it is possible to significantly reduce the dose of Remifentanil, in order to avoid episodes of respiratory depression caused by the opioid.

The secondary outcomes measured, will be the pain levels experienced by the patient, the sedation level, and the satisfaction of the patients after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients having an oocyte retrieval

Exclusion Criteria:

* BMI > 30
* endometriosis
* contraindications to ketamine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients in good health, with informed consent, undergoing oocyte retrieval at the Erasmus Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
respiratory depression | through study completion, an average of 2 months
  respiratory rate (number of inspiration per minute)
Respiratory depression | through study completion, an average of 2 months
  SpO2 (%)

SECONDARY OUTCOMES:
pain | through study completion, an average of 2 months
  EVA
patient satisfaction | through study completion, an average of 2 months
  satisfaction scale: 1=unsatisfied. 2=average satisfaction 3=Satisfied 4=very satisfied. The higher the value, the better. Additionally, we ask the patients if they would choose the same anesthetic method, should it be necessary to repeat the procedure. If yes, it is considered a better outcome.
pregnancy rate | 15 days after the oocyte retrieval
  HCG in the blood
ketamine dosage | through study completion, an average of 2 months
  blood sample (serum)
sedation level | through study completion, an average of 2 months
  OAAS: Observer's Assessment Of Alertness/Sedation Scale. 5=Responds readily to name spoken in normal tone. 4=Lethargic response to name spoken in normal tone. 3=Response only after name is called loudly and/or repeatedly. 2=Response only after mild prodding or shaking. 1=Response only after paintful trapezius squeeze. 0=No response after paintful trapezius squeeze. Values higher than 3 represents a better outcome.
Arterial pressure | through study completion, an average of 2 months
  mmHg
Heart rate | through study completion, an average of 2 months
  Beats per minute
Pain | through study completion, an average of 2 months
  NOL-index
Pain | through study completion, an average of 2 months
  ANI
Sedation level | through study completion, an average of 2 months
  Ramsay sedation scale. 1=Anxious and agitated or restless, or both. 2=Co-operative, oriented, and calm. 3=Responsive to commands only. 4=Exhibiting brisk response to light glabellar tap or loud auditory stimulus. 5=Exhibiting a sluggish response to light glabellar tap or loud auditory stimulus. 6=unresponsive. Values of 2-3 represent the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peres-Bota Iulia, student, Principal Investigator — Erasme University Hospital; Barvais Luc, MDPhD, Study Director — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Belgium